CLINICAL TRIAL: NCT05333055
Title: Aqueous Biomarker Levels in Diabetic Retinopathy and Diabetic Macular Edema
Acronym: DRAGONS
Status: Terminated | Type: Observational
Why Stopped: Dissolution of the ophthalmology department
Sponsor: Greater Houston Retina Research (Other)
Responsible Party: Sponsor
Other Study IDs: DRAGONS
Record Dates: First submitted 2022-04-11; First posted 2022-04-18 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-09

CONDITIONS: Diabetic Retinopathy; Diabetic Macular Edema; Other Retinal Disorders
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Aqueous humor, plasma and serum will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group 1: Eyes with treatment naive DR with or without DME
- Group 2: Eyes with DME that are incompletely responsive to anti-VEGF therapy
- Group 3: Eyes with various retinal conditions including eyes with DR and DME that is anti-VEGF responsive as well as non-exudative retinal pathologies such as epiretinal membrane and macular hole

SUMMARY:
The DRAGONS study is a non-interventional, prospective study that will

1. characterize disease state biomarker (including cytokines, KKS metabolites, and cell adhesion molecules) levels from aqueous humor of subjects with various stages of diabetic retinopathy (DR) and diabetic macular edema (DME) as well as other retinal pathologies, and
2. correlate a broad array of aqueous humor disease state biomarkers with DR severity, DME anti-vascular endothelial growth factor (VEGF) responsiveness, and other retinal pathologies.

DETAILED DESCRIPTION:
The DRAGONS study is a non-interventional study investigating aqueous humor biomarker levels in patients with various stages of DR, DME and other retinal pathologies.

Subjects will be included in the study if at least one eye meets any of the following criteria:

Group 1 - eyes with treatment naive DR with or without DME Group 2 - eyes with DME that are incompletely responsive to anti-VEGF therapy Group 3 - eyes with various retinal conditions including eyes with DR and DME that are anti-VEGF responsive as well as non-exudative retinal pathologies such as epiretinal membrane and macular hole

The study will consist of a single visit and a retrospective chart review. The study visit will consist of:

1. Screening for eligibility;
2. Aqueous humor collection;
3. Blood collection;
4. Optical coherence tomography;
5. Optical coherence tomography angiography;
6. Fundus photography; and
7. Fluorescein angiography.

Approximately 50 microliters (or more, up to 150 microliters) of aqueous fluid will be collected according to standard clinical procedures. Plasma and serum will be collected according to standard clinical procedures, with citrated plasma being specifically collected in a plastic tube.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with at least one of the following retinal conditions in at least one eye:

* Treatment naive diabetic retinopathy (group 1 only);
* Diabetic retinopathy with DME that is incompletely responsive to anti-VEGF therapy at principal investigators discretion with retinal thickening documented on OCT (group 2 only);
* Various retinal disease including but not limited to diabetic retinopathy without DME which has previously been treated, DME which has responded to anti-VEGF therapy, neovascular age-related macular degeneration, branch or central retinal vein occlusions, epiretinal membrane, or macular hole (group 3 only)

Exclusion Criteria:

1. Prior intraocular or subtenon steroid injection in the study eye within the prior 1 year of signing informed consent;
2. Prior focal or grid laser photocoagulation in the study eye if within 90 days of signing informed consent;
3. Prior panretinal photocoagulation in the study eye if within 90 days of signing informed consent;
4. Intraocular or refractive surgery in the study eye within 90 days of signing informed consent;
5. Systemic anti-VEGF treatment within 90 days of signing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retina Consultants of Texas patient population
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Aqueous Humor Levels of Disease State Biomarkers | Baseline
  Aqueous humor levels of cytokines, KKS metabolites, and cell adhesion molecules of subjects with various stages of diabetic retinopathy and diabetic macular edema as well as other retinal pathologies.

SECONDARY OUTCOMES:
Correlation of Biomarker Levels | Baseline
  Correlation of aqueous humor disease state biomarkers with diabetic retinopathy severity, diabetic macular edema anti-VEGF responsiveness, and other retinal pathologies.

CONTACTS AND LOCATIONS:
Overall Officials: Charles C. Wykoff, MD, PhD, Principal Investigator — Greater Houston Retina Research
Locations (3):
- United States (3):
  - Retina Consultants of Texas, Bellaire, Texas
  - Retina Consultants of Texas, Katy, Texas
  - Retina Consultants of Texas, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kempen JH, O'Colmain BJ, Leske MC, Haffner SM, Klein R, Moss SE, Taylor HR, Hamman RF; Eye Diseases Prevalence Research Group. The prevalence of diabetic retinopathy among adults in the United States. Arch Ophthalmol. 2004 Apr;122(4):552-63. doi: 10.1001/archopht.122.4.552. PMID 15078674
- [Background] Leasher JL, Bourne RR, Flaxman SR, Jonas JB, Keeffe J, Naidoo K, Pesudovs K, Price H, White RA, Wong TY, Resnikoff S, Taylor HR; Vision Loss Expert Group of the Global Burden of Disease Study. Global Estimates on the Number of People Blind or Visually Impaired by Diabetic Retinopathy: A Meta-analysis From 1990 to 2010. Diabetes Care. 2016 Sep;39(9):1643-9. doi: 10.2337/dc15-2171. PMID 27555623
- [Background] Bourne RR, Stevens GA, White RA, Smith JL, Flaxman SR, Price H, Jonas JB, Keeffe J, Leasher J, Naidoo K, Pesudovs K, Resnikoff S, Taylor HR; Vision Loss Expert Group. Causes of vision loss worldwide, 1990-2010: a systematic analysis. Lancet Glob Health. 2013 Dec;1(6):e339-49. doi: 10.1016/S2214-109X(13)70113-X. Epub 2013 Nov 11. PMID 25104599
- [Background] Aiello LP, Avery RL, Arrigg PG, Keyt BA, Jampel HD, Shah ST, Pasquale LR, Thieme H, Iwamoto MA, Park JE, et al. Vascular endothelial growth factor in ocular fluid of patients with diabetic retinopathy and other retinal disorders. N Engl J Med. 1994 Dec 1;331(22):1480-7. doi: 10.1056/NEJM199412013312203. PMID 7526212
- [Background] Mesquida M, Drawnel F, Fauser S. The role of inflammation in diabetic eye disease. Semin Immunopathol. 2019 Jul;41(4):427-445. doi: 10.1007/s00281-019-00750-7. Epub 2019 Jun 7. PMID 31175392
- [Background] Mesquita J, Castro-de-Sousa JP, Vaz-Pereira S, Neves A, Passarinha LA, Tomaz CT. Evaluation of the growth factors VEGF-a and VEGF-B in the vitreous and serum of patients with macular and retinal vascular diseases. Growth Factors. 2018 Apr;36(1-2):48-57. doi: 10.1080/08977194.2018.1477140. Epub 2018 Jul 3. PMID 29969324
- [Background] Amadio M, Govoni S, Pascale A. Targeting VEGF in eye neovascularization: What's new?: A comprehensive review on current therapies and oligonucleotide-based interventions under development. Pharmacol Res. 2016 Jan;103:253-69. doi: 10.1016/j.phrs.2015.11.027. Epub 2015 Dec 8. PMID 26678602
- [Background] Witmer AN, Vrensen GF, Van Noorden CJ, Schlingemann RO. Vascular endothelial growth factors and angiogenesis in eye disease. Prog Retin Eye Res. 2003 Jan;22(1):1-29. doi: 10.1016/s1350-9462(02)00043-5. PMID 12597922
- [Background] Zhang X, Bao S, Lai D, Rapkins RW, Gillies MC. Intravitreal triamcinolone acetonide inhibits breakdown of the blood-retinal barrier through differential regulation of VEGF-A and its receptors in early diabetic rat retinas. Diabetes. 2008 Apr;57(4):1026-33. doi: 10.2337/db07-0982. Epub 2008 Jan 3. PMID 18174522
- [Background] Hofman P, Blaauwgeers HG, Tolentino MJ, Adamis AP, Nunes Cardozo BJ, Vrensen GF, Schlingemann RO. VEGF-A induced hyperpermeability of blood-retinal barrier endothelium in vivo is predominantly associated with pinocytotic vesicular transport and not with formation of fenestrations. Vascular endothelial growth factor-A. Curr Eye Res. 2000 Aug;21(2):637-45. PMID 11148600
- [Background] Early photocoagulation for diabetic retinopathy. ETDRS report number 9. Early Treatment Diabetic Retinopathy Study Research Group. Ophthalmology. 1991 May;98(5 Suppl):766-85. PMID 2062512
- [Background] Photocoagulation treatment of proliferative diabetic retinopathy. Clinical application of Diabetic Retinopathy Study (DRS) findings, DRS Report Number 8. The Diabetic Retinopathy Study Research Group. Ophthalmology. 1981 Jul;88(7):583-600. PMID 7196564
- [Background] Diabetic Retinopathy Clinical Research Network; Elman MJ, Aiello LP, Beck RW, Bressler NM, Bressler SB, Edwards AR, Ferris FL 3rd, Friedman SM, Glassman AR, Miller KM, Scott IU, Stockdale CR, Sun JK. Randomized trial evaluating ranibizumab plus prompt or deferred laser or triamcinolone plus prompt laser for diabetic macular edema. Ophthalmology. 2010 Jun;117(6):1064-1077.e35. doi: 10.1016/j.ophtha.2010.02.031. Epub 2010 Apr 28. PMID 20427088
- [Background] Nguyen QD, Brown DM, Marcus DM, Boyer DS, Patel S, Feiner L, Gibson A, Sy J, Rundle AC, Hopkins JJ, Rubio RG, Ehrlich JS; RISE and RIDE Research Group. Ranibizumab for diabetic macular edema: results from 2 phase III randomized trials: RISE and RIDE. Ophthalmology. 2012 Apr;119(4):789-801. doi: 10.1016/j.ophtha.2011.12.039. Epub 2012 Feb 11. PMID 22330964
- [Background] Korobelnik JF, Do DV, Schmidt-Erfurth U, Boyer DS, Holz FG, Heier JS, Midena E, Kaiser PK, Terasaki H, Marcus DM, Nguyen QD, Jaffe GJ, Slakter JS, Simader C, Soo Y, Schmelter T, Yancopoulos GD, Stahl N, Vitti R, Berliner AJ, Zeitz O, Metzig C, Brown DM. Intravitreal aflibercept for diabetic macular edema. Ophthalmology. 2014 Nov;121(11):2247-54. doi: 10.1016/j.ophtha.2014.05.006. Epub 2014 Jul 8. PMID 25012934
- [Background] Fong DS, Girach A, Boney A. Visual side effects of successful scatter laser photocoagulation surgery for proliferative diabetic retinopathy: a literature review. Retina. 2007 Sep;27(7):816-24. doi: 10.1097/IAE.0b013e318042d32c. PMID 17891003
- [Background] Ferris F. Early photocoagulation in patients with either type I or type II diabetes. Trans Am Ophthalmol Soc. 1996;94:505-37. PMID 8981711
- [Background] Writing Committee for the Diabetic Retinopathy Clinical Research Network; Gross JG, Glassman AR, Jampol LM, Inusah S, Aiello LP, Antoszyk AN, Baker CW, Berger BB, Bressler NM, Browning D, Elman MJ, Ferris FL 3rd, Friedman SM, Marcus DM, Melia M, Stockdale CR, Sun JK, Beck RW. Panretinal Photocoagulation vs Intravitreous Ranibizumab for Proliferative Diabetic Retinopathy: A Randomized Clinical Trial. JAMA. 2015 Nov 24;314(20):2137-2146. doi: 10.1001/jama.2015.15217. PMID 26565927
- [Background] Bolinger MT, Antonetti DA. Moving Past Anti-VEGF: Novel Therapies for Treating Diabetic Retinopathy. Int J Mol Sci. 2016 Sep 7;17(9):1498. doi: 10.3390/ijms17091498. PMID 27618014
- [Background] Stitt AW, Curtis TM, Chen M, Medina RJ, McKay GJ, Jenkins A, Gardiner TA, Lyons TJ, Hammes HP, Simo R, Lois N. The progress in understanding and treatment of diabetic retinopathy. Prog Retin Eye Res. 2016 Mar;51:156-86. doi: 10.1016/j.preteyeres.2015.08.001. Epub 2015 Aug 18. PMID 26297071
- [Background] Stewart MW. Treatment of diabetic retinopathy: Recent advances and unresolved challenges. World J Diabetes. 2016 Aug 25;7(16):333-41. doi: 10.4239/wjd.v7.i16.333. PMID 27625747
- [Background] Maturi RK, Bleau L, Saunders J, Mubasher M, Stewart MW. A 12-MONTH, SINGLE-MASKED, RANDOMIZED CONTROLLED STUDY OF EYES WITH PERSISTENT DIABETIC MACULAR EDEMA AFTER MULTIPLE ANTI-VEGF INJECTIONS TO ASSESS THE EFFICACY OF THE DEXAMETHASONE-DELAYED DELIVERY SYSTEM AS AN ADJUNCT TO BEVACIZUMAB COMPARED WITH CONTINUED BEVACIZUMAB MONOTHERAPY. Retina. 2015 Aug;35(8):1604-14. doi: 10.1097/IAE.0000000000000533. PMID 25829346
- [Background] Wu H, Hwang DK, Song X, Tao Y. Association between Aqueous Cytokines and Diabetic Retinopathy Stage. J Ophthalmol. 2017;2017:9402198. doi: 10.1155/2017/9402198. Epub 2017 Jun 7. PMID 28680705
- [Background] Dong N, Xu B, Wang B, Chu L. Study of 27 aqueous humor cytokines in patients with type 2 diabetes with or without retinopathy. Mol Vis. 2013 Aug 4;19:1734-46. Print 2013. PMID 23922491
- See also: 2016 Global Report on Diabetes — http://apps.who.int/iris/bitstream/10665/204871/1/9789241565257_eng.pdf?ua=1&ua=1.